CLINICAL TRIAL: NCT02013466
Title: Amino Acid Bioavailability in Healthy Elderly After Bolus Intake of a High Whey-protein, Leucine-rich, Low-caloric Oral Nutritional Supplement
Brief Title: Amino Acid Bioavailability in Healthy Elderly After Intake of an Oral Nutritional Supplement
Acronym: ArenA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Sip.1.C/B
Record Dates: First submitted 2013-12-02; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Sarcopenia
Keywords: Bioavailability; Amino Acids; Elderly; Supplement
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bolus ONS intake (Other): Bolus ONS A Bolus ONS B Bolus ONS C Bolus ONS D ONS = oral nutritional supplement 4-way cross-over design: Determination of the product order is based on a Latin square design. 3 Latin squares (4x4) are used, resulting in 12 unique product orders. Subjects receive a randomisation number corresponding with 1 of the 12 product orders. Study product labels will contain randomisation number and appropriate visit number.
  Interventions: Dietary Supplement: Bolus ONS A; Dietary Supplement: Bolus ONS B; Dietary Supplement: Bolus ONS C; Dietary Supplement: Bolus ONS D

INTERVENTIONS:
Dietary Supplement: Bolus ONS A — High-whey protein, leucine-rich, low-caloric ONS in powder format
Dietary Supplement: Bolus ONS B — High casein-protein, low-caloric control product (isocaloric to product A)
Dietary Supplement: Bolus ONS C — High casein-protein, high-caloric control product.
Dietary Supplement: Bolus ONS D — high whey-protein, leucine-rich, high-caloric control product (isocaloric to product C)

SUMMARY:
In this study healthy older adults are requested to consume 4 different high-protein nutritional supplements. Each subject will visit the site 4 times and at every visit they will consume 1 of the 4 products after which a series of blood samples will be taken. The blood samples will be analyzed for amino acid bioavailability in the blood up to 4 hours after consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* BMI between 21 and 30 kg/m2

Exclusion Criteria:

* Any condition that may interfere with the definition 'healthy elderly' according to the investigator's judgement.
* Any (history of) gastrointestinal disease that interferes with GI function (e.g. inflammatory bowel disease, gastroparesis, gastrectomy).
* Known allergy to milk and milk products.
* Known galactosaemia.
* Current or recent (within past three months) smoking.
* Known or suspected Diabetes Mellitus.
* Current infection or fever in the last 7 days at the discretion of the physician.
* Use of antibiotics within 3 weeks of study entry.
* Current use of corticosteroids or hormones.
* Current use of antacids or any medication influencing gastric acid production.
* Requirement for any nutritional support.
* Unplanned body weight loss > 5% in the past 3-6 months.
* Adherence to any specific diet (e.g. weight loss, vegetarian).
* Use of protein containing or amino acid containing nutritional supplements within one week of study entry.
* Alcohol or drug abuse.
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.
* Participation in any other study with investigational products concomitantly or within 4 weeks of study entry.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome parameter in this study is the Maximum serum leucine concentration (Leumax) [micromol/L]. | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)

SECONDARY OUTCOMES:
Serum leucine incremental area under the curve (iAUC) [micromol/L*min]. | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Time to reach half the serum leucine iAUC (t½) [minutes]. | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Maximum serum essential amino acid concentration (EAAmax) [micromol/L] | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Maximum serum amino acid concentration (AAmax) [mmol/L] | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Maximum serum insulin concentration [micromol/L]. | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Serum insulin iAUC [micromol/L*min] | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Maximum serum glucose concentration [mmol/L] | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Serum glucose iAUC [mmol/L*min] | Up to 4 hours after each bolus intake (4 visits, 7-10 days between 2 consecutive visits)
Adverse events and (Gastro-Intestinal) tolerance questionnaire. | During the study and until one week after completion of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Ampha, Nijmegen, Netherlands

REFERENCES:
- [Derived] Luiking YC, Abrahamse E, Ludwig T, Boirie Y, Verlaan S. Protein type and caloric density of protein supplements modulate postprandial amino acid profile through changes in gastrointestinal behaviour: A randomized trial. Clin Nutr. 2016 Feb;35(1):48-58. doi: 10.1016/j.clnu.2015.02.013. Epub 2015 Mar 5. PMID 25790724